CLINICAL TRIAL: NCT03178071
Title: AN EXPANDED ACCESS PROTOCOL FOR LORLATINIB FOR TREATMENT OF PATIENTS WITH ADVANCED NON-SMALL CELL LUNG CANCER HARBORING SPECIFIC MOLECULAR ALTERATIONS
Brief Title: Expanded Access For Lorlatinib For Patients With Non Small Cell Lung Cancer ALK Positive or ROS1 Positive
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461020
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Non Small Cell Lung Cancer ALK Positive or ROS1 Positive
Keywords: NSCLC
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Lorlatinib — oral tablets, administered daily, continuously
  Other Names: PF-06463922

SUMMARY:
This expanded access study has being designed following a demand from the FDA, given the increase in the number of request for single patient INDs for lorlatinib

DETAILED DESCRIPTION:
Given that an Expanded Access study does not meet the definition of a controlled clinical investigation, and as such, is not considered an applicable drug clinical trial per NIH, Basic Results for such studies are not required to be reported. Protocol B7461020 has been identified as an Expanded Access trial, and has been registered to ClinicalTrials.gov, however Basic Results will not be posted. This statement has been placed in the Detailed Description section of the protocol registration on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Ineligibility for participation in any ongoing clinical study of the investigational product
* Age ≥18 years
* Histologically or cytologically diagnosis of metastatic NSCLC that carries an ALK rearrangement or a ROS1 rearrangement
* For ALK positive patients: failure to prior treatment with at least one ALK-TKI. If prior ALK-TKI was crizotinib, additional prior treatment required with at least one second generation ALK-TKI registered and commercially available. For patients with resistance mutations not covered by other inhibitors (eg, ALK G1202R resistance mutation), prior treatment with an ALK/ROS1 inhibitor is not required.
* For ROS1 positive patients: failure to prior treatment with at least crizotinib
* Adequate bone marrow, liver, renal, pancreatic functions
* Negative pregnancy test at screening

Exclusion Criteria:

* Previous surgery, chemotherapy, radiotherapy or other anti cancer therapy or participation in other studies with investigational drugs within the timeframe indicated in the protocol
* History of interstitial fibrosis or interstitial lung disease
* Concomitant use of prohibited medication
* Clinically significant cardiovascular disease: cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure, second degree or third degree atrioventricular block (unless paced) or any AV block with PR >220 msec
* Ongoing cardiac dysrhythmias, uncontrolled atrial fibrillation,bradycardia, ECG with QTc >470 msec, or congenital long QT syndrome
* History of or predisposing characteristics for acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- United States (47):
  - Arizona Oncology Associates, PC - NAHOA, Sedona, Arizona
  - Pacific Shores Medical Group, Huntington Beach, California
  - Pacific Shores Medical Group, Irvine, California
  - Pacific Shores Medical Group, Long Beach, California
  - Kaiser Permanente, Oakland Medical Center, Oakland, California
  - UC Irvine Health / Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Irvine/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente, South Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente, San Francisco Medical Center, San Francisco, California
  - Kaiser Permanente, Vallejo Medical Center, Vallejo, California
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - University Cancer & Blood Center, Llc, Athens, Georgia
  - University of Chicago Medical Center, CCD, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Elmhurst Memorial Hospital Nancy W. Knowles Cancer Center, Elmhurst, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute/Pharmacy, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Rutgers Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Breast and Imaging Center - 12th floor, New York, New York
  - North Shore Hematology Oncology Associates, Patchogue, New York
  - North Shore Hematology Oncology Associates, Port Jefferson Station, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University East Hospital, Columbus, Ohio
  - The Ohio State University Investigational Drug Services, Columbus, Ohio
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - The Ohio State University Martha Morehouse Medical Plaza, Columbus, Ohio
  - CarePoint Gahanna, Gahanna, Ohio
  - UPMC Hillman Cancer Center - Patient Clinic, Pittsburgh, Pennsylvania
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461020